CLINICAL TRIAL: NCT05623982
Title: An Open, Multicenter, Phase Ib/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of Tetra-specific Antibody GNC-038 Injection in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma (NHL)
Brief Title: A Study of GNC-038 Injection in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry); Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GNC-038-104
Record Dates: First submitted 2022-08-25; First posted 2022-11-21 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Non-hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive GNC-038 as intravenous infusion for the first cycle (2 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: GNC-038

INTERVENTIONS:
Drug: GNC-038 — Administration by intravenous infusion

SUMMARY:
To explore the safety and preliminary efficacy of GNC-038 in patients with relapsed or refractory NHL, and to determine the MTD and RP2D of GNC-038, or the MAD and DLT

DETAILED DESCRIPTION:
phase Ib: To explore the safety and preliminary efficacy of GNC-038 in patients with relapsed or refractory NHL, and to determine the MTD and RP2Dof GNC-038, or the MAD and DLT of GNC-038 if MTD is not reached, by intravenous infusion (IV, QW) once a week (2 weeks as a cycle) phase II To explore the efficacy of GNC-038 in patients with relapsed or refractory non-Hodgkin's lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. The subject is capable of understanding the informed consent form, voluntarily participates, and signs the informed consent form;
2. No gender restrictions;
3. Age: ≥18 years and ≤75 years;
4. Expected survival time ≥3 months;
5. Patients with histologically confirmed non-Hodgkin's lymphoma;
6. Patients with relapsed or refractory non-Hodgkin's lymphoma (R/R NHL);
7. Presence of measurable lesions during the screening period (lymph node lesions with any long diameter ≥1.5 cm or extranodal lesions with any long diameter >1.0 cm);
8. ECOG performance status score ≤2;
9. Adverse reactions from prior anti-tumor treatment have recovered to ≤Grade 1 as per CTCAE 5.0 criteria;
10. Organ function levels meet the requirements before the first dose;
11. Female subjects of childbearing potential or male subjects with partners of childbearing potential must use highly effective contraception from 7 days before the first dose until 12 weeks after treatment discontinuation. Female subjects of childbearing potential must have a negative serum/urine pregnancy test within 7 days before the first dose;
12. The subject has the ability and willingness to comply with the study protocol-specified visits, treatment plans, laboratory tests, and other study-related procedures.

Exclusion Criteria:

1. Pulmonary diseases classified as ≥Grade 3 according to NCI-CTCAE v5.0; patients currently diagnosed with interstitial lung disease (ILD);
2. Active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.;
3. Active tuberculosis;
4. Patients with active autoimmune diseases;
5. History of other malignancies within 5 years prior to the first dose;
6. HBsAg-positive and/or HBcAb-positive with HBV-DNA levels ≥ the lower limit of detection; HCV antibody-positive with HCV-RNA levels ≥ the lower limit of detection; HIV antibody-positive;
7. Poorly controlled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg);
8. History of severe cardiovascular or cerebrovascular diseases;
9. Patients with a history of hypersensitivity to recombinant humanized antibodies or any excipients of GNC-038;
10. Pregnant or lactating women;
11. Patients with central nervous system involvement;
12. Major surgery within 28 days before the first dose of this study or planned major surgery during the study period;
13. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
14. Autologous hematopoietic stem cell transplantation (Auto-HSCT) within 12 weeks before initiating GNC-038 treatment;
15. Current use of immunosuppressive therapy;
16. Radiotherapy within 4 weeks before initiating GNC-038 treatment;
17. Chemotherapy or small-molecule targeted therapy within 2 weeks or 5 half-lives prior to treatment;
18. CAR-T therapy within 12 weeks before initiating GNC-038 treatment;
19. Use of any other investigational drug in a clinical trial within 4 weeks or 5 half-lives before the first dose of this study;
20. Any other condition deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 14 days after the first dose
  The incidence and severity of adverse events (TEAE) during treatment were graded according to the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI-CTCAE, v5.0).
Maximum tolerated dose (MTD) or Maximum dose (MAD) | Up to 14 days after the first dose
  In the dose increment stage, the highest dose whose estimated DLT rate is closest to the target DLT rate but does not exceed the upper bound of the equivalent interval of DLT rate is selected as MTD.
Adverse Events during Treatment (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-038. The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-038.
Recommended dose for Phase II clinical studies (RP2D) | Up to 14 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of GNC-038.

SECONDARY OUTCOMES:
disease control rate (DCR) | Up to approximately 24 months
  Number of patients showing Complete Response (CR) or Partial Response (PR) based on RECIST for the best response.
  Number of patients showing Complete Response (CR, disappearance of all target lesions) or Partial Response (PR, at least a 30% decrease in the sum of longest diameter of target lesions taking as reference the baseline sum longest diameter) based on RECIST Criteria Version 1.0 (assessed by CT and/or MRI) for the best response.
progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of GNC-038 to the first date of either disease progression or death, whichever occurs first.
Adverse Events of Special Interest (AESI) | Up to approximately 24 months
  AESI is an event of scientific and medical interest specific to the sponsor's product or research project.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of GNC-038 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of GNC-038 will be investigated.
AUC0-INF | Up to approximately 24 months
  Blood concentration - Area under time line.
AUC0-T | Up to approximately 24 months
  Blood concentration - Area under time line.
T1/2 | Up to approximately 24 months
  Blood concentration - Area under time line.
anti-drug antibody (ADA) in Ⅰa | Up to approximately 24 months
  Frequency and titer of anti-GNC-038 antibody (ADA).
DOR (Duration of Response) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.

OTHER OUTCOMES:
Neutralizing antibody (Nab) in phase Ⅰb | Up to approximately 24 months
  Incidence and titer of Nab of GNC-038 will be evaluated.
Overall survival (OS) in phaseⅠb and phase Ⅱ | Up to approximately 24 months
  The time between the start of study medication and death.
Neutralizing antibody (Nab) in phaseⅡ | Up to approximately 24 months
  Incidence and titer of Nab of GNC-038 will be evaluated.
anti-drug antibody (ADA) in phaseⅡ | Up to approximately 24 months
  Frequency and titer of anti-GNC-038 antibody (ADA) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, Principal Investigator — Peking University Cancer Hospital & Institute; Yuqin Song, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Harbin First Hospital, Haerbin, Heilongjing
  - Qingdao Central Hospital, Qingdao, Shandong

IPD SHARING:
Plan to Share IPD: No